CLINICAL TRIAL: NCT02287168
Title: Effect of Peritoneal Lavage on Surgery-induced Positive Peritoneal Cytology in Gastric Cancer Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Mustafa Hasbahceci, MD, general surgeon, Bezmialem Vakif University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GastCancPerLav2014
Record Dates: First submitted 2014-10-31; First posted 2014-11-10 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Gastric Adenocarcinoma; Gastric Cancer
Keywords: Peritoneal lavage; Dissemination; Gastrectomy; Cytology; Lavage
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- dissemination of cancer cells (Experimental): conversion of negative result of pre-gastrectomy peritoneal washing cytology to positive cytology after gastrectomy
  Interventions: Procedure: pre-gastrectomy peritoneal washing cytology; Procedure: post-gastrectomy peritoneal washing cytology
- elimination of cancer cells (Experimental): elimination of peritoneal cancer cells occurred before (pre-gastrectomy peritoneal washing cytology) or after gastrectomy (post-gastrectomy peritoneal washing cytology) by intra operative peritoneal lavage ('post-lavage peritoneal washing cytology)
  Interventions: Procedure: pre-gastrectomy peritoneal washing cytology; Procedure: post-gastrectomy peritoneal washing cytology; Procedure: post-lavage peritoneal washing cytology

INTERVENTIONS:
Procedure: pre-gastrectomy peritoneal washing cytology — sampling of peritoneal washing fluid before gastrectomy
Procedure: post-gastrectomy peritoneal washing cytology — sampling of peritoneal washing fluid after gastrectomy
Procedure: post-lavage peritoneal washing cytology — sampling of peritoneal washing fluid after peritoneal lavage
  Arms: elimination of cancer cells

SUMMARY:
Surgical manipulation and handling of a tumor may cause dissemination of cancer cells through peritoneal cavity after curative gastrectomy. Intra operative peritoneal lavage may have preventive effect on positive peritoneal cytology occurred during gastrectomy in patients with gastric cancer.

DETAILED DESCRIPTION:
Peritoneal dissemination of gastric adenocarcinoma cells is the most frequent cause of death in patients with gastric cancer. Spreading of these cells occur by three routes: direct seeding via infiltration through gastric wall, via blood vessels and via perigastric lymphatic channels disturbed during lymph node dissection. Conversion of negative preoperative peritoneal cytology to positive cytology after curative gastrectomy has been shown by previous studies.

Although extensive intra-operative peritoneal lavage (1 L of physiologic saline 10 times) has been shown to be an effective method to eliminate cancer cell dissemination during surgery, to cause significant improvement in survival after gastrectomy, widespread use of this approach has not existed most probably due to its time consuming technical difficulty. Therefore,intra-operative peritoneal lavage (1 L of physiologic saline 3 times) may be used more frequently during gastric surgery.If it is possible to show effectivity of intra-operative peritoneal lavage using a total of 3 L physiologic saline to eliminate cancer cell dissemination occurred before or after gastric surgery, use of this approach may gain acceptance to decrease risk of peritoneal metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopically proven gastric adenocarcinoma
* Standard gastrectomy and a D2 lymph node dissection;
* Desire to attend the study protocol

Exclusion Criteria:

* Metastatic or overt peritoneal disseminated cancer
* Undesired reaction to attend the study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
elimination | at the operation
  rate of conversion of positive cytology results to negative cytology by peritoneal lavage during the surgery

SECONDARY OUTCOMES:
dissemination | at the operation
  rate of conversion of negative cytology results to positive cytology by surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Bezmialem Vakif University Faculty of Medicine Dept of General Surgery, Istanbul
  - Mustafa Hasbahceci, Istanbul

REFERENCES:
- [Background] Yu XF, Ren ZG, Xue YW, Song HT, Wei YZ, Li CM. D2 lymphadenectomy can disseminate tumor cells into peritoneal cavity in patients with advanced gastric cancer. Neoplasma. 2013;60(2):174-81. doi: 10.4149/neo_2013_023. PMID 23259786
- [Background] Shimada S, Kuramoto M, Marutsuka T, Yagi Y, Baba H. Adopting extensive intra-operative peritoneal lavage (EIPL) as the standard prophylactic strategy for peritoneal recurrence. Rev Recent Clin Trials. 2011 Sep;6(3):266-70. doi: 10.2174/157488711796575603. PMID 21682671
- [Background] Yamamoto K, Shimada S, Hirota M, Yagi Y, Matsuda M, Baba H. EIPL (extensive intraoperative peritoneal lavage) therapy significantly reduces peritoneal recurrence after pancreatectomy in patients with pancreatic cancer. Int J Oncol. 2005 Nov;27(5):1321-8. PMID 16211228
- [Background] Misawa K, Mochizuki Y, Ohashi N, Matsui T, Nakayama H, Tsuboi K, Sakai M, Ito S, Morita S, Kodera Y. A randomized phase III trial exploring the prognostic value of extensive intraoperative peritoneal lavage in addition to standard treatment for resectable advanced gastric cancer: CCOG 1102 study. Jpn J Clin Oncol. 2014 Jan;44(1):101-3. doi: 10.1093/jjco/hyt157. Epub 2013 Nov 27. PMID 24287077
- [Background] Kuramoto M, Shimada S, Ikeshima S, Matsuo A, Yagi Y, Matsuda M, Yonemura Y, Baba H. Extensive intraoperative peritoneal lavage as a standard prophylactic strategy for peritoneal recurrence in patients with gastric carcinoma. Ann Surg. 2009 Aug;250(2):242-6. doi: 10.1097/SLA.0b013e3181b0c80e. PMID 19638909
- [Background] Marutsuka T, Shimada S, Shiomori K, Hayashi N, Yagi Y, Yamane T, Ogawa M. Mechanisms of peritoneal metastasis after operation for non-serosa-invasive gastric carcinoma: an ultrarapid detection system for intraperitoneal free cancer cells and a prophylactic strategy for peritoneal metastasis. Clin Cancer Res. 2003 Feb;9(2):678-85. PMID 12576435
- [Background] Shimada S, Tanaka E, Marutsuka T, Honmyo U, Tokunaga H, Yagi Y, Aoki N, Ogawa M. Extensive intraoperative peritoneal lavage and chemotherapy for gastric cancer patients with peritoneal free cancer cells. Gastric Cancer. 2002;5(3):168-72. doi: 10.1007/s101200200029. PMID 12378344